CLINICAL TRIAL: NCT03127852
Title: Randomized Controlled Trial of a Mobile Phone-based Telemonitoring Application for Self-management and Clinical Decision Support for Patients With Complex Chronic Conditions
Brief Title: Effects of Remote Patient Monitoring on Chronic Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-9995
Record Dates: First submitted 2016-08-09; First posted 2017-04-25 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease; Chronic Kidney Disease; Uncontrolled Hypertension; Diabetes
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Renal Insufficiency, Chronic; Diabetes Mellitus

ARMS (2):
- Telemonitoring (Medly) (Experimental): The telemonitoring technology will enable patients with complex chronic illnesses, to take clinically relevant physiological measurements with wireless home medical devices and to answer symptom questions on the mobile phone. The measurements will be automatically and wirelessly transmitted to the mobile phone and then to a data server. Automated self-care instructions/messages will be sent to the patient based on the readings and reported symptoms. If there are signs of their status deteriorating, an alert will be sent to a clinician that is responsible for the particular chronic condition of concern. The clinicians will have all the relevant patient data sent to them and will be able to access (through a secure web portal) to view historical and trending data for their patients.
  Interventions: Device: Medly
- Control (No Intervention): Standard of care: Patients are followed in a specialty care clinic treating their primary conditions. Patients typically have scheduled appointments every six months.

INTERVENTIONS:
Device: Medly
  Arms: Telemonitoring (Medly)

SUMMARY:
Remote patient monitoring is a potential component for the management of chronic conditions that may provide reliable and real-time physiological measurements for clinical decision support, alerting, and patient self-management. The purpose of this study is to evaluate an UHN-built remote monitoring system for patients with complex chronic conditions called Medly.

DETAILED DESCRIPTION:
Remote patient monitoring is a potential component for the management of chronic conditions that may provide reliable and real-time physiological measurements for clinical decision support, alerting, and patient self-management. The purpose of this study is to evaluate an UHN-built remote monitoring system for patients with complex chronic conditions called Medly. Patients with complex chronic conditions will be provided with a mobile phone and commercial home medical devices, such as a blood pressure monitor and weight scale. The measurements from the medical devices will be automatically sent to the mobile phone, and from there to a data server at the hospital for analysis and storage. Both clinicians and patients will be able to access these data and will be sent alerts by the system if the measurements are outside of the normal range. The system will be evaluated through interviews and comparing outcomes between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. Adults (age 18 years or older)
2. Diagnosed with HF, COPD, CKD, and/or uncontrolled hypertension (individuals with diabetes who require blood glucose monitoring will be included as a co-morbidity only if patient's have at least one of the above four chronic illnesses, and will be in the form of self-care support only)
3. Patient or their caregiver speaks and reads English adequately to provide informed consent and understand the text prompts in the application.
4. Ability to comply with using the telemonitoring system (e.g, able to stand on the weight scale, able to answer symptom questions, etc.).

Primary chronic disease-specific criteria:

* Patients with HF as the primary chronic disease: with reduced ejection fraction (EF<0.40)
* Patients with COPD as the primary chronic disease: Spirometrically confirmed diagnosis of COPD of GOLD Stage II or higher (defined as post-bronchodilator FEV1 < 80% predicted and FEV1/FVC ratio < 70%); smoking history of ≥ 20 pack-years or homozygous alpha-1 antitrypsin deficiency; and prescribed an action plan for the early self-treatment of acute exacerbations
* Patients with CKD as the primary chronic disease: Grade 3-5 (eGFR < 60mL/1.73 m2)
* Patients with uncontrolled hypertension as the primary chronic disease: For non-diabetics: blood pressure >=140/90 mmHg auscultatory (manual measurement) or >=135/85 mmHg oscillometric (automated measurement). For diabetics: blood pressure >=130/80 mmHg

Exclusion Criteria:

1. Patients on mechanical circulatory support
2. Patients on the heart transplant list
3. Terminal diagnosis with life expectancy < 1 year
4. Dementia or uncontrolled psychiatric illness
5. Resident of a long term care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ware P, Shah A, Ross HJ, Logan AG, Segal P, Cafazzo JA, Szacun-Shimizu K, Resnick M, Vattaparambil T, Seto E. Challenges of Telemonitoring Programs for Complex Chronic Conditions: Randomized Controlled Trial With an Embedded Qualitative Study. J Med Internet Res. 2022 Jan 26;24(1):e31754. doi: 10.2196/31754. PMID 35080502
- [Derived] Seto E, Ware P, Logan AG, Cafazzo JA, Chapman KR, Segal P, Ross HJ. Self-Management and Clinical Decision Support for Patients With Complex Chronic Conditions Through the Use of Smartphone-Based Telemonitoring: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2017 Nov 21;6(11):e229. doi: 10.2196/resprot.8367. PMID 29162557

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemonitoring (Medly): The telemonitoring technology will enable patients with complex chronic illnesses, to take clinically relevant physiological measurements with wireless home medical devices and to answer symptom questions on the mobile phone. The measurements will be automatically and wirelessly transmitted to the mobile phone and then to a data server. Automated self-care instructions/messages will be sent to the patient based on the readings and reported symptoms. If there are signs of their status deteriorating, an alert will be sent to a clinician that is responsible for the particular chronic condition of concern. The clinicians will have all the relevant patient data sent to them and will be able to access (through a secure web portal) to view historical and trending data for their patients.
  Medly
Period: Overall Study
Arm/Group | Telemonitoring (Medly) | Control
Started | 46 | 50
Completed | 41 | 48
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemonitoring (Medly) | Control | Total
Number analyzed (Participants) | 46 | 50 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12.6) | 55 (14.3) | 59 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Participants
    number analyzed (Participants) | 37 | 34 | 71
    Female | 9 | 8 | 17
    Male | 28 | 26 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Number analyzed reflects the number of participants who provided responses to this question.
  Participants
    White: number analyzed (Participants) | 34 | 36 | 70
    White | 22 | 24 | 46
    Black: number analyzed (Participants) | 34 | 36 | 70
    Black | 2 | 4 | 6
    Asian: number analyzed (Participants) | 34 | 36 | 70
    Asian | 3 | 6 | 9
    Other: number analyzed (Participants) | 34 | 36 | 70
    Other | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 46 | 50 | 96
Highest Education Achieved [Count of Participants; unit: Participants] — Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Participants
    number analyzed (Participants) | 34 | 35 | 69
    Less than high school | 4 | 1 | 5
    High school | 5 | 4 | 9
    Trade or technical training | 5 | 6 | 11
    College or university | 15 | 19 | 34
    Postgraduate | 5 | 5 | 10
Comfort with Smartphone [Count of Participants; unit: Participants] — Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Participants
    number analyzed (Participants) | 30 | 47 | 77
    Not comfortable | 1 | 0 | 1
    Somewhat comfortable | 8 | 4 | 12
    Comfortable | 8 | 28 | 36
    Very comfortable | 13 | 15 | 28
SF-36 (Physical Component) [Mean (Standard Deviation); unit: units on a scale] — 36-Item Short Form Survey (SF-36) measures health-related quality of life. It consists of 2 component summary measures: physical and mental health. The Physical Component Summary (PCS) measure is derived from domain scales of Physical Functioning (10 items), Role-Physical (4 items), Bodily Pain (2 items), and General Health (5 items). Component summary measure scores range from 0 to 100 with higher scores indicating better outcomes. Norm-based scoring was used so that scores for each component summary measure has a mean of 50 (standardized to the US population) and standard deviation of 10. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 24 | 25 | 49
    (all) | 40.94 (8.11) | 41.55 (8.86) | 41.25 (8.42)
SF-36 (Mental Component) [Mean (Standard Deviation); unit: units on a scale] — 36-Item Short Form Survey (SF-36) measures health-related quality of life and consists of 2 component summary measures: physical and mental health. The Mental Component Summary (MCS) measure is derived from domain scales of: Vitality (4 items), Social Functioning (2 items), Role-emotional (3 items), and Mental Health (5 items). Component summary measure scores range from 0 to 100 with higher scores indicating better outcomes. Norm-based scoring was used so that scores for each component summary measure has a mean of 50 (standardized to the US population) and standard deviation of 10. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 24 | 25 | 49
    (all) | 46.42 (12.21) | 46.96 (11.21) | 46.70 (11.59)
HADS (Anxiety) [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS) has two sub-scales for anxiety and depression. Scores for items in the anxiety sub-scale are summed to produce an anxiety score (HADS-A). The anxiety sub-scale has scores ranging from 0 to 21, with higher scores indicating higher levels of anxiety Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 24 | 22 | 46
    (all) | 6.94 (4.38) | 6 (4) | 6.49 (4.18)
HADS (Depression) [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS) has two sub-scales for anxiety and depression. Scores for items in the depression sub-scale are summed to produce a depression score (HADS-D). The depression sub-scale has scores ranging from 0 to 21, with higher scores indicating higher levels of depression. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 5.09 (3.95) | 5.21 (3.85) | 5.15 (3.86)
SEMCD6 [Mean (Standard Deviation); unit: units on a scale] — Each item on the Self-Efficacy for Managing Chronic Disease 6-Item scale (SEMCD6) is rated from 1 (not at all confident) to 10 (totally confident). The final score for the scale is the mean of the six items with higher scores indicating higher self-efficacy. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 26 | 24 | 50
    (all) | 7.23 (2.18) | 7.08 (2.55) | 7.16 (2.34)
Hospital visits [Mean (Standard Deviation); unit: Visits] — Self-reported number of hospital visits Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Visits
    number analyzed (Participants) | 28 | 23 | 51
    (all) | 4.29 (10.56) | 3.7 (6.51) | 4.02 (8.89)
ED visits [Mean (Standard Deviation); unit: Visits] — Self-reported emergency department visits Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Visits
    number analyzed (Participants) | 28 | 23 | 51
    (all) | 1.29 (4.65) | 0.071 (1.34) | 0.74 (3.58)
Clinic visits [Mean (Standard Deviation); unit: Visits] — Self-reported clinic visits Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Visits
    number analyzed (Participants) | 20 | 21 | 41
    (all) | 3.54 (4.11) | 4.19 (6.01) | 3.87 (5.12)
Family physician visits [Mean (Standard Deviation); unit: Visits] — Self-reported family physician visits Population: Number analyzed reflects the number of participants who returned the baseline survey.
  Visits
    number analyzed (Participants) | 25 | 23 | 48
    (all) | 1.65 (1.22) | 2.48 (3.72) | 2.05 (2.72)
SCHFI (Maintenance) [Mean (Standard Deviation); unit: units on a scale] — Self-Care of Heart Failure Index (SCHFI) has three scales: maintenance, management, confidence. The self-care maintenance subscale includes 10 items asking how often patients check their heart failure symptoms and treatment adherence. The score is standardized to a 0- to 100-point range with each scale score standardized to a 0 to 100 range with 0 indicating the worst and 100 indicating the best performance for each scale score. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 24 | 17 | 41
    (all) | 73.42 (14.77) | 73.64 (15.75) | 73.51 (14.99)
SCHFI (Management) [Mean (Standard Deviation); unit: units on a scale] — Self-Care of Heart Failure Index (SCHFI) has three scales: maintenance, management, confidence. The self-care management sub-scale includes 6 items if patients report any heart failure symptoms in the past month. Then based on the responses on how quick they recognize it as a symptom of heart failure and remedies they tried. The score is standardized to a 0- to 100-point range with each scale score standardized to a 0 to 100 range with 0 indicating the worst and 100 indicating the best performance for each scale score. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 24 | 17 | 41
    (all) | 71.75 (15.64) | 64.47 (27.51) | 68.73 (21.37)
SCHFI (Confidence) [Mean (Standard Deviation); unit: units on a scale] — Self-Care of Heart Failure Index (SCHFI) has three scales: maintenance, management, confidence. The self-care confidence subscale includes 6 items asking how confident that they can keep themselves free of symptoms, follow treatment advice, recognize changes in their health and etc. The score is standardized to a 0- to 100-point range with each scale score standardized to a 0 to 100 range with 0 indicating the worst and 100 indicating the best performance for each scale score. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 24 | 16 | 40
    (all) | 69.43 (15.49) | 69.94 (25.09) | 69.63 (19.59)
MLHFQ (Total) [Mean (Standard Deviation); unit: units on a scale] — Minnesota Living with Heart Failure Questionnaire (MLHFQ) provides a total score which ranges from 0-105. A lower total score is indicative of better quality of life. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 23 | 17 | 40
    (all) | 40.85 (28.52) | 42.81 (26.15) | 41.68 (27.21)
MLHFQ (Physical) [Mean (Standard Deviation); unit: units on a scale] — Minnesota Living with Heart Failure Questionnaire (MLHFQ) provides a total score, as well as scores for two dimensions, physical and emotional. The sum of points of the physical dimension sub-scale (8 items) ranges from 0-40 and a lower physical score is indicative of better quality of life. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 23 | 17 | 40
    (all) | 19.13 (11.01) | 20.78 (10.64) | 19.83 (10.75)
MLHFQ (Emotional) [Mean (Standard Deviation); unit: units on a scale] — Minnesota Living with Heart Failure Questionnaire (MLHFQ) provides a total score, as well as scores for two dimensions, physical and emotional. The sum of points of the emotional dimension sub-scale (5 items) ranges from 0-25 and a lower emotional score is indicative of better quality of life. Population: Number analyzed reflects the number of participants who returned the baseline survey.
  units on a scale
    number analyzed (Participants) | 22 | 15 | 37
    (all) | 10.38 (7.97) | 11.38 (7.08) | 10.79 (7.54)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life as Measured by SF-36
Description: Change in Quality of life as measured by the Short Form (36) Health Survey. The SF-36 assesses participants' overall quality of life in eight domains 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 contribute to the physical component summary (PCS) score, and items 5-8 contribute to the mental component summary (MCS) score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemonitoring (Medly) | Control
Number analyzed (Participants) | 24 | 25
score on a scale
  Physical Component | 42.77 (8.58) | 42.39 (9.47)
  Mental Component | 43.77 (12.28) | 48.31 (10.51)
Statistical Analysis 1: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of SF-36 physical component summary score; Test type: Superiority; p = .48, t-test, 2 sided
Statistical Analysis 2: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of SF-36 mental component summary score; Test type: Superiority; p = .73, t-test, 2 sided

2. Secondary Outcome: Self-reported Health Service Use
Description: Number of hospitalizations, number of ED and clinic visits, and family physician visits.
Time Frame: Baseline, 6 months
Population: Number of participants analyzed reflects those who completed the follow-up survey. Shifting priorities at the onset of the COVID-19 pandemic affected the collection of poststudy data, as patients followed for hypertension and diabetes mellitus ended their enrollment during the first wave of the pandemic, which led to a higher rate of incomplete questionnaires.
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Telemonitoring (Medly) | Control
Number analyzed (Participants) | 28 | 23
Visits
  Hospital (number of visits) | 1.43 (4.11) | 0.35 (1.11)
  ED visits | 0.5 (1.33) | 0.22 (0.57)
  Clinic visits: number analyzed (Participants) | 20 | 21
  Clinic visits | 3.71 (2.85) | 2.95 (4.61)
  Family physician visits: number analyzed (Participants) | 25 | 23
  Family physician visits | 1.28 (1.62) | 1.85 (2.23)
Statistical Analysis 1: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of self-reported number of hospital visits; Test type: Superiority; p = .02, t-test, 2 sided
Statistical Analysis 2: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of self-reported emergency department visits; Test type: Superiority; p = .12, t-test, 2 sided
Statistical Analysis 3: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of self-reported number of clinic visits; Test type: Superiority; p = .39, t-test, 2 sided
Statistical Analysis 4: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of self-reported number of family physician visits; Test type: Superiority; p = .28, t-test, 2 sided

3. Secondary Outcome: Self-Care of Health Failure as Measured by the SCHFI
Description: Self-care of health failure as measured by the Self-Care of Heart Failure Index (SCHFI). The SCFHI has three scales: maintenance, management, confidence with each scale score is standardized to a 0 to 100 range with 0 indicating the worst and 100 indicating the best performance for each scale score.
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemonitoring (Medly) | Control
Number analyzed (Participants) | 24 | 17
score on a scale
  Maintenance | 79.83 (15.81) | 76.18 (17.48)
  Management | 75.42 (19.83) | 69.53 (26.53)
  Confidence: number analyzed (Participants) | 24 | 16
  Confidence | 71.83 (19.74) | 76.38 (19.86)
Statistical Analysis 1: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of SCHFI maintenance sub-scale; Test type: Superiority; p = .74, t-test, 2 sided
Statistical Analysis 2: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of SCHFI management sub-scale; Test type: Superiority; p = .67, t-test, 2 sided
Statistical Analysis 3: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of SCHFI confidence sub-scale; Test type: Superiority; p = .92, t-test, 2 sided

4. Secondary Outcome: Heart-failure Specific Quality of Life (MLHFQ)
Description: Heart-failure specific quality of life as measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The MLHFQ provides a total score (score range 0-105), as well as scores for two dimensions, physical (score range 0-40) and emotional (score range 0-25). A lower total score is indicative of better quality of life.
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemonitoring (Medly) | Control
Number analyzed (Participants) | 23 | 17
score on a scale
  Total | 35.88 (23.65) | 31.55 (29.45)
  Physical | 14.58 (10.9) | 19.05 (12.4)
  Emotional: number analyzed (Participants) | 22 | 15
  Emotional | 9 (7.45) | 9.33 (7.1)
Statistical Analysis 1: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of MLHFQ total score; Test type: Superiority; p = .67, t-test, 2 sided
Statistical Analysis 2: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of MLHFQ physical domain score; Test type: Superiority; p = .43, t-test, 2 sided
Statistical Analysis 3: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of MLHFQ emotional domain score; Test type: Superiority; p = .64, t-test, 2 sided

5. Secondary Outcome: Anxiety and Depression as Measured by HADS
Description: Anxiety and depression as measured by the Hospital Anxiety and Depression Scale (HADS). The HADS has two sub-scales for anxiety and depression. Each sub-scale has scores ranging from 0 to 21, with higher scores indicating higher levels of anxiety/depression.
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemonitoring (Medly) | Control
Number analyzed (Participants) | 24 | 23
score on a scale
  Anxiety | 7.33 (5.07) | 5.97 (3.5)
  Depression | 5.51 (4.67) | 5.55 (4.2)
Statistical Analysis 1: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of HADS anxiety sub-scale; Test type: Superiority; p = .06, t-test, 2 sided
Statistical Analysis 2: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of HADS depression sub-scale; Test type: Superiority; p = .77, t-test, 2 sided

6. Secondary Outcome: Self-efficacy as Measured by the SEMCD6.
Description: Self-efficacy as measured by the Self-Efficacy for Managing Chronic Disease 6-Item scale (SEMCD6). Each item on the scale is rated from 1 (not at all confident) to 10 (totally confident). The final score for the scale is the mean of the six items with higher scores indicating higher self-efficacy.
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemonitoring (Medly) | Control
Number analyzed (Participants) | 26 | 24
score on a scale | 7.35 (1.57) | 6.75 (2.21)
Statistical Analysis 1: Comparison: Telemonitoring (Medly) vs Control; Poststudy between-group comparison of SEMCD6; Test type: Superiority; p = .13, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Telemonitoring (Medly) | Control
All-Cause Mortality (participants affected / at risk) | 1/46 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/50
Other Adverse Events (participants affected / at risk) | 0/46 | 0/50

LIMITATIONS AND CAVEATS:
Early termination of recruitment before reaching the target sample size because (1) the HF telemonitoring program became standard of care; (2) recruitment challenges observed for patients with DM because of the rapid emergence and growing use of continuous and flash glucose monitors; and (3) the COVID-19 pandemic led to a pause of nonessential research activities and a significant shift toward virtual care, which fundamentally altered the control group after the research pause was lifted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03127852/Prot_SAP_000.pdf